CLINICAL TRIAL: NCT00002977
Title: A Phase I Trial of Melphalan and Thiotepa Followed by Autologous or Syngeneic Peripheral Blood Stem Cell (PBSC) Rescue in Patients With a Complete Response Following Standard Therapy for Stage III/IV Epithelial Ovarian Cancer
Brief Title: Melphalan and Thiotepa Followed by Peripheral Stem Cell Transplantation in Treating Patients With Epithelial Ovarian Cancer in Complete Remission
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1181.00; 1181.00; NCI-G97-1229; CDR0000065499 (Registry Identifier: PDQ)
Record Dates: First submitted 1999-11-01; First posted 2004-04-29 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2010-09

CONDITIONS: Ovarian Cancer
Keywords: stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; recurrent ovarian epithelial cancer; ovarian undifferentiated adenocarcinoma; ovarian mixed epithelial carcinoma; ovarian serous cystadenocarcinoma; ovarian mucinous cystadenocarcinoma; ovarian endometrioid adenocarcinoma; ovarian clear cell cystadenocarcinoma; Brenner tumor
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial; Brenner Tumor | interventions — Filgrastim; Melphalan; Thiotepa; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: filgrastim
Drug: melphalan
Drug: thiotepa
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of melphalan and thiotepa followed by peripheral stem cell transplantation in treating patients with stage III or stage IV epithelial ovarian cancer in complete remission.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the toxic effects of combined high dose melphalan and thiotepa chemotherapy followed by stem cell rescue in patients with stage III or IV ovarian epithelial cancer in complete remission. II. Determine the maximum tolerated dose of thiotepa that can be given with melphalan in these patients. III. Evaluate the interpatient blood level variability and pharmacokinetics of melphalan given intravenously.

OUTLINE: This is a dose escalation study of thiotepa. Patients receive cytoreduction and mobilization of peripheral blood stem cells (PBSC) with filgrastim (G-CSF) and cyclophosphamide/paclitaxel, cyclophosphamide/etoposide or cyclophosphamide/etoposide/cisplatin within 30-90 days of last dose of standard therapy. PBSC are then collected. Patients then receive melphalan IV over 30 minutes on days -6 and -5 and thiotepa IV over 2 hours on days -4 and -3. PBSC are reinfused on day 0. G-CSF is administered on days 0-21. Cohorts of 5-15 patients each receive escalating doses of thiotepa until the maximum tolerated dose (MTD) is reached. The MTD is determined as the dose at which 2-5 of 4-15 patients experience dose limiting toxicity. Patients are followed at 100 days, then at 6, 12, and 24 months.

PROJECTED ACCRUAL: A total of 30-45 patients will be accrued for this study over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed stage III/IV ovarian epithelial cancer in first or second clinical complete remission after receiving a minimum of 4-10 courses of chemotherapy consisting of paclitaxel and either cisplatin or carboplatin Ovarian epithelial cancer of following histologic types: Serous adenocarcinoma Mucinous adenocarcinoma Clear cell adenocarcinoma Transitional cell Adenocarcinoma N.O.S. Endometrioid adenocarcinoma Undifferentiated carcinoma Mixed epithelial carcinoma Malignant Brenner's Tumor Remission stability maintained for at least 4 weeks Protocol therapy must begin 30-90 days after last dose of standard therapy No active pleural or pericardial effusion No prior/concurrent brain metastasis or carcinoid meningitis

PATIENT CHARACTERISTICS: Age: 18 to 60 Performance status: Karnofsky 70-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Bilirubin less than 1.5 times the upper limit of normal (ULN) SGOT or SGPT less than 2.0 times ULN Albumin greater than 2.0 g/dL Renal: Creatinine clearance greater than 60 mL/min Cardiovascular: Ejection fraction greater than 45% by MUGA Pulmonary: If history of smoking or abnormal lung function, Diffusion capacity greater than 50% (corrected) A-a gradient less than 20 Other: No history of hemorrhagic cystitis No second malignancy within the last 5 years except basal cell skin cancer HIV negative No chronic active hepatitis B No hepatitis C No history of Aspergillus infection

PRIOR CONCURRENT THERAPY: Biologic therapy: No prior stem cell transplant Chemotherapy: Prior chemotherapy consisting of paclitaxel and either cisplatin or carboplatin Endocrine therapy: Not specified Radiotherapy: No prior radiation therapy for malignancy (excluding chest wall radiation therapy for breast cancer) Surgery: Not specified

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 1997-01; Primary Completion 2001-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leona A. Holmberg, MD, PhD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States